CLINICAL TRIAL: NCT07229599
Title: A Phase I/II Clinical Study to Evaluate the Efficacy and Safety of MHB036C for Injection Combined With Other Anti-tumor Therapy in Patients With Advanced Lung Cancer
Brief Title: A Study of MHB036C Combined With Anti-tumor Therapies in Patients With Advanced Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MHB036C-A-201
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lung Cancer
MeSH Terms: interventions — Injections; aflutinib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose escalation: cohort 1 (Experimental): Subjects will receive MHB036C Q3W by intravenous administration in combination with Furmonertinib QD by oral administration.
  Interventions: Drug: MHB036C for Injection; Drug: Furmonertinib
- Dose escalation: cohort 2 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Dose escalation: cohort 3 (Experimental): Subjects will receive MHB036C Q3W in combination with Carboplatin AUC 5mg/mL/min by intravenous administration
  Interventions: Drug: MHB036C for Injection; Drug: Carboplatin
- Dose expansion: cohort 4 (Experimental): Subjects will receive MHB036C Q3W by intravenous administration in combination with Furmonertinib QD by oral administration.
  Interventions: Drug: MHB036C for Injection; Drug: Furmonertinib
- Dose expansion: cohort 5 (Experimental): Subjects will receive MHB036C Q3W in combination with MHB039A Q3W by intravenous administration
  Interventions: Drug: MHB036C for Injection; Drug: MHB039A for Injection
- Dose expansion: cohort 6 (Experimental): Subjects will receive MHB036C Q3W in combination with Carboplatin AUC 5mg/mL/min by intravenous administration
  Interventions: Drug: MHB036C for Injection; Drug: Carboplatin

INTERVENTIONS:
Drug: MHB036C for Injection — IV administration; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
Drug: MHB039A for Injection — IV administration; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
  Arms: Dose escalation: cohort 2; Dose expansion: cohort 5
Drug: Furmonertinib — Oral administration; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
  Arms: Dose escalation: cohort 1; Dose expansion: cohort 4
Drug: Carboplatin — IV administration; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.
  Arms: Dose escalation: cohort 3; Dose expansion: cohort 6

SUMMARY:
This is a first-in-human, open-label, multicenter Phase I/II study of MHB036C combined with MHB039A or other anti-tumor therapy in patients with advanced lung cancer. The study was designed to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of MHB036C combined with MHB039A or other anti-tumor therapies.

DETAILED DESCRIPTION:
This first-in-human clinical trial of MHB036C combined with MHB039A or other anti-tumor therapy comprises two parts: a dose escalation phase and dose expansion phase. The dose escalation phase is an open-label, multicenter study including dose escalation and PK expansion cohorts. The primary objectives are to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of MHB036C combining different anti-tumor treatment regimens (including Furmonertinib, MHB039A for injection, and Carboplatin) in patients with advanced lung cancer, and to determine the maximum tolerated dose (MTD). Additional patients may be enrolled in the PK expansion part at dose levels that have completed DLT (dose-limiting toxicity) evaluation.

Based on the safety, PK, and preliminary efficacy data from the completed DLT-evaluated dose levels, the sponsor will initiate the dose expansion phase to further evaluate the safety and efficacy of MHB036C combined with MHB039A or other anti-tumor therapy in patients with specific types of advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agrees to participate in the study and signs the informed consent form.
2. Age ≥ 18 years and≤75 years, no restriction on gender.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Estimated life expectancy ≥ 3 months.
5. For the dose escalation stage: Histologically or cytologically confirmed advanced solid tumors that are refractory to standard therapy, intolerant to standard therapy, or have no standard treatment options.
6. For the dose expansion stage: Histologically or cytologically confirmed locally advanced or metastatic advanced solid tumors, not suitable for radical surgery and/or radical concurrent/sequential radiotherapy and chemotherapy.
7. At least one measurable lesion per RECIST v1.1 criteria.
8. Adequate bone marrow reserve and organ function.
9. Eligible participants of childbearing potential (males and females) must agree to take highly reliable contraceptive measures with their partners during the study and within at least 12 weeks after the last dose.

   -

Exclusion Criteria:

1. Small cell lung cancer (SCLC) components in the histopathology.
2. History of ≥2 primary malignancies within 5 years prior to informed consent.
3. Received chemotherapy within 3 weeks, radiotherapy within 4 weeks, or biologic, endocrine, or immunotherapy within 4 weeks before first study dose.
4. Medication of other unmarketed investigational drugs or therapies within 4 weeks before dosing.
5. Brain metastases, leptomeningeal disease, brainstem metastases, or spinal cord compression.
6. Underwent major organ surgery (excluding biopsy) or significant trauma within 4 weeks before the first dose of investigational drug or requiring elective surgery during the study.
7. Previous or concurrent gastrointestinal perforation, surgical procedures and wound healing complications, as well as bleeding events.
8. Received intravenous thrombolysis treatment within 2 weeks, except for preventive anticoagulation and antiplatelet therapy.
9. Vaccinated within 4 weeks before dosing.
10. Treated with systemic corticosteroids within 14 days before dosing.
11. Severe impairment of pulmonary function; interstitial lung disease or a history of pneumonia requiring steroid treatment; previous left or right pneumonectomy.
12. Active systemic infection requiring treatment within 7 days before dosing.
13. Uncontrolled third-space effusion.
14. Serious cardiovascular or cerebrovascular diseases.
15. Known hypersensitivity or delayed allergic reaction to the investigational product or its components.
16. Drug abuse or other medical/psychiatric condition that may interfere with study participation or results.
17. Known alcohol or drug dependence.
18. Pregnant or breastfeeding women, or individuals planning to conceive. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
(Dose-Escalation Stage): Maximum tolerated dose (MTD) for MHB036C and other anti-tumor treatment combination therapy | Up to day 21 from the first dose for Q3W administration.
  To determine the MTD for further evaluation of MHB036C and other anti-tumor treatment combination therapy
(Dose-Escalation Stage): Incidence and severity of adverse events (AEs) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years.
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0].
(Dose-Expansion Stage): Objective tumor response (ORR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat).

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of total antibody, ADC, and free toxin at various time points | From pre-dose to 22 days after the first dose
  The PK parameters at different time points include: Area Under the Concentration-Time Curve (AUC)
Pharmacokinetic (PK) parameters of total antibody, ADC, and free toxin at various time points | From pre-dose to 22 days after the first dose
  The PK parameters at different time points include: Maximum Plasma Concentration (Cmax)
Duration of response (DOR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Disease control rate (DCR) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose].
Progression-free survival (PFS) determined by investigators according to RECIST v1.1 | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 5 years
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). PFS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to PD or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No